CLINICAL TRIAL: NCT03928197
Title: Discovering the Effect of Venous Insufficiency on Nocturia (DEVINe - Trial) - Pilootstudie: definiëren Van Duidelijke Afkapwaarden Omtrent Oedeem Ter Hoogte Van de Onderste Ledematen te Gevolge Van Veneuze insufficiëntie.
Brief Title: Discovering the Effect of Venous Insufficiency on Nocturia (DEVINe)
Acronym: DEVINe Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UZG 2019/0022
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Edema Leg; Venous Insufficiency of Leg; Nocturia; Bio-Impedance Measurements
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Other)
  Interventions: Behavioral: Tilt Test; Device: Inbody S10; Device: Tape measurements; Device: SOMNOtouchTMNIBP, Vivisol, Belgium
- Volunteers with Venous Insuficiency (Other)
  Interventions: Behavioral: Tilt Test; Device: Inbody S10; Device: Tape measurements; Device: SOMNOtouchTMNIBP, Vivisol, Belgium

INTERVENTIONS:
Behavioral: Tilt Test — Volunteers need to lay down for 15 minutes and afterwards stand up for 15 minutes
Device: Inbody S10 — Bio-electrical impedance measurement every 5 minutes
Device: Tape measurements — Every 5 minutes, circumference of every leg is measured using a tape measure
Device: SOMNOtouchTMNIBP, Vivisol, Belgium — Continous measurement of blood pressure, heart rate and saturation

SUMMARY:
Nocturia, or waking during the night to pass urine, is a multifactorial disease. An important cause of nocturia are peripheral edema due to accumulation of fluid in the lower limbs. Venous insufficiency is an important cause of peripheral edema. The investigators hypothesize that, as a result of the lying position during the night, the accumulated fluid in the lower limbs returns to the systemical circulation leading and is excreted during nighttime. This will lead to a higher voiding frequency during the night.

With this trail the investigators wanst to prove the difference in leg edema between healthy volunteers and volunteers with venous insufficiency (Type 1 or 2).

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 years and 60 years
* For the volunteers with venous insuffiency: clearly visual venous insufficiency (CEAP 1 and 2)
* BMI between 24 and 30

Exclusion Criteria:

* Volunteers using medication (exception for contraception)
* Volunteers having comorbidities
* Pregnant women
* Women who menstruate on the test date
* Volunteers with an implanted elektronical device (IPG, Pacemaker)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Leg swelling measured in cm | 25 minutes
  Difference in lower limb swelling between healthy volunteers and volunteers with venous insufficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided